CLINICAL TRIAL: NCT03136536
Title: Kärlkirurgi Vid Komplicerade kroppspulsåderbråck - Utfall, Riskfaktorer Och sökande Efter biomarkörer för Organskada
Brief Title: Organ Failure After Advanced Endovascular Thoracoabdominal Aortic Surgery
Acronym: ODEA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 206471
Record Dates: First submitted 2017-04-19; First posted 2017-05-02 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Aortic Aneurysm; Spinal Ischaemia; Gastrointestinal Ischaemia
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, urine, cerebrospinal fluid, intraperitoneal microdialysate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the mortality and frequency of organ dysfunction in patients after endovascular thoracoabdominal aortic surgery, and to search for biomarkers of organ dysfunction, in particular the spinal cord, the kidneys and the gastrointestinal tract. All adult patients undergoing endovascular thoracoabdominal aortic surgery at Örebro University Hospital, Örebro, Sweden, are asked for participation in this study. All participating patients sign informed consent at the inclusion. During the operation and during the postoperative intensive care, the function of the spinal cord, the gastrointestinal tract and the kidneys are collected along with other clinical parameters. Plasma blood samples, urin samples and cerebrospinal fluid samples are collected from each patient during the operation and during the postoperative care at the intensive care unit. During the operation two microdialysis catheters are placed in the abdomen, and the samples are continuously collected and analyzed. The biomaterial samples are stored in a biobank for later determination of proteins and other molecules. Postoperative survival and the frequency of complications are analysed.

ELIGIBILITY:
Inclusion Criteria:

* Accepted for endovascular advanced thoracoabdominal aortic surgical procedure
* Adult

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing endovascular advanced thoracoabdominal aortic surgical procedures at Örebro University Hospital, Örebro, Sweden.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year postoperative
  Overall and aortic-related mortality

SECONDARY OUTCOMES:
Organ dysfunction and failure | Postoperative: 7 days, 30 days, 1 year follow-up
  Spinal cord, gastrointestinal tract, kidneys

OTHER OUTCOMES:
Proteomics | Postoperative: 7 days
  Plasma, urine, cerebrospinal fluid, intraperitoneal microdialysate

CONTACTS AND LOCATIONS:
Overall Officials: Kristofer F Nilsson, MD, PhD, Principal Investigator — Department of Cardio-thoracic and Vascular Surgery, Faculty of Medicine and Health, Örebro University, Örebro, Sweden
Locations (1):
- Department of Cardio-thoracic and Vascular Surgery, Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No